CLINICAL TRIAL: NCT03171116
Title: Unacylated Ghrelin and Obestatin as Promising Biomarkers of Protein Energy Wasting in Children With Chronic Kidney Disease: a Cross-sectional Case-control Study
Brief Title: Ghrelin and Obestatin in CKD Children
Status: Completed | Type: Observational
Sponsor: Azienda Ospedaliero Universitaria Maggiore della Carita (Other)
Responsible Party: Principal Investigator, Flavia Prodam, Clinical Professor, Azienda Ospedaliero Universitaria Maggiore della Carita
Other Study IDs: 396/2011 bis
Record Dates: First submitted 2017-05-25; First posted 2017-05-31 (Actual); Last update posted 2017-05-31 (Actual); Status verified 2017-05

CONDITIONS: Chronic Kidney Diseases
Keywords: ghrelin; obestatin; children
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- CKD-CT: subjects with CKD stages II-V under conservative treatment
  Interventions: Other: none intervention
- CKD-HD: subjects with CKD stage V on hemodialysis
  Interventions: Other: none intervention
- RTx renal transplant: renal transplant recipients
  Interventions: Other: none intervention
- Controls: control subjects
  Interventions: Other: none intervention

INTERVENTIONS:
Other: none intervention — it is not an interventional study; it is an observational study

SUMMARY:
Protein energy wasting (PEW) is a complex syndrome associated with different underlying illnesses and characterized by loss of muscle, with or without loss of fat. It is a highly prevalent condition among patients with chronic kidney disease (CKD), associated with increased morbidity and mortality.

The pathophysiology of PEW in CKD is multifactorial and not yet completely understood. The potential role in uremic PEW of two of hormones involved in orexigenic/anorexigenic balance, ghrelin and obestatin, both derived from the ghrelin gene (GHRL), has been investigated in adults and, less extensively, in children. Aim of our study was to measure AG, UAG and obestatin concentrations in children with CKD and to assess their potential contribution to the development of pediatric uremic PEW.

DETAILED DESCRIPTION:
This is a cross-sectional case-control study. Between January 2013 and June 2015 children and adolescents aged 5-20 years, referred to the Pediatric Nephrology, Dialysis and Transplant Unit of Fondazione IRCCS Ca' Granda - Ospedale Maggiore Policlinico - Milan, Italy were enrolled. Subjects with CKD stages II-V under conservative treatment (CKD-CT), or undergoing hemodialysis treatment (CKD-HD), or being renal transplant recipients (RTx) were included in the study. Data about age, primary renal disease and concomitant medications were collected for each subject.

CKD stages were defined using the K/DOQI criteria of the US National Kidney Foundation.

Control subjects were outpatients of the Pediatric Surgery Unit of the Fondazione IRCCS Ca' Granda - Ospedale Maggiore Policlinico - Milan, Italy, aged 1-20 years, who underwent a blood sample collection before a surgical intervention for the treatment of minor diseases that did not impair renal or endocrine function (i.e. phimosis, hydrocele, inguinal hernia).

Biochemical and hormonal parameters Blood samples were collected between 7:00 and 8:00 a.m. after an overnight fast, and before dialysis in CKD-HD patients. Routine biochemical parameters [creatinine, urea] were measured in all subjects. Glomerular filtration rate was estimated (eGFR) by the Schwartz formula, with k = 0.413, as appropriate for standardized creatinine.

In all subjects, plasma AG and UAG concentrations were measured by the Human Acylated / Unacylated Ghrelin ELISA kit (BioVendor, Laboratorni Medicina a.s., Brno, Czech Republic) according to manufacture procedures, and AG/UAG ratio was calculated. Serum obestatin concentrations were determined using the Human Obestatin ELISA kit (BioVendor, Laboratorni Medicina a.s., Brno, Czech Republic).

ELIGIBILITY:
Inclusion Criteria:

* the CKD-HD patients should have been on hemodialysis treatment for at least 3 months
* the RTx patients should have received renal transplantation at least 6 months before

Exclusion Criteria:

* treatment with growth hormone
* the presence of neurologic disability or syndromic diseases affecting per se food intake
* for controls: they should have no history of chronic diseases and should not receive any medication. They should be on unrestricted diet.

Ages: 5 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: A total of 154 subjects were included (M:F=100:54), 111 patients and 43 controls. Out of 111 patients, 43 had CKD stages II-V under conservative treatment (CKD-CT), 20 were on hemodialysis (CKD-HD), 48 were renal transplant recipients (RTx).
Sampling Method: Probability Sample
Enrollment: 154 (Actual)
Dates: Start 2013-01-01 (Actual); Primary Completion 2015-06-30 (Actual); Study Completion 2015-06-30 (Actual)

PRIMARY OUTCOMES:
AG concentrations by ELISA kit on plasma samples | January 2013-June 2015
  Acyl-ghrelin measurement
UAG concentrations by ELISA kit on plasma samples | January 2013-June 2015
  Unacyl-ghrelin measurement
Obestatin concentrations by ELISA kit on serum samples | January 2013-June 2015
  Obestatin measurement

CONTACTS AND LOCATIONS:
Overall Officials: Flavia Prodam, MD, Study Director — Università del Piemonte Orientale - Novara

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mak RH, Ikizler AT, Kovesdy CP, Raj DS, Stenvinkel P, Kalantar-Zadeh K. Wasting in chronic kidney disease. J Cachexia Sarcopenia Muscle. 2011 Mar;2(1):9-25. doi: 10.1007/s13539-011-0019-5. Epub 2011 Mar 16. PMID 21475675
- [Background] Perez-Fontan M, Cordido F, Rodriguez-Carmona A, Peteiro J, Garcia-Naveiro R, Garcia-Buela J. Plasma ghrelin levels in patients undergoing haemodialysis and peritoneal dialysis. Nephrol Dial Transplant. 2004 Aug;19(8):2095-100. doi: 10.1093/ndt/gfh313. Epub 2004 Jun 8. PMID 15187192
- [Background] Iglesias P, Diez JJ, Fernandez-Reyes MJ, Codoceo R, Alvarez-Fidalgo P, Bajo MA, Aguilera A, Selgas R. Serum ghrelin concentrations in patients with chronic renal failure undergoing dialysis. Clin Endocrinol (Oxf). 2006 Jan;64(1):68-73. doi: 10.1111/j.1365-2265.2005.02418.x. PMID 16402931
- [Background] Barazzoni R, Zanetti M, Stulle M, Mucci MP, Pirulli A, Dore F, Panzetta G, Vasile A, Biolo G, Guarnieri G. Higher total ghrelin levels are associated with higher insulin-mediated glucose disposal in non-diabetic maintenance hemodialysis patients. Clin Nutr. 2008 Feb;27(1):142-9. doi: 10.1016/j.clnu.2007.06.013. Epub 2007 Sep 12. PMID 17854954
- [Background] Jarkovska Z, Hodkova M, Sazamova M, Rosicka M, Dusilova-Sulkova S, Marek J, Justova V, Lacinova Z, Haluzik M, Haas T, Krsek M. Plasma levels of active and total ghrelin in renal failure: a relationship with GH/IGF-I axis. Growth Horm IGF Res. 2005 Dec;15(6):369-76. doi: 10.1016/j.ghir.2005.07.004. Epub 2005 Sep 28. PMID 16198134
- [Background] Yoshimoto A, Mori K, Sugawara A, Mukoyama M, Yahata K, Suganami T, Takaya K, Hosoda H, Kojima M, Kangawa K, Nakao K. Plasma ghrelin and desacyl ghrelin concentrations in renal failure. J Am Soc Nephrol. 2002 Nov;13(11):2748-52. doi: 10.1097/01.asn.0000032420.12455.74. PMID 12397045
- [Background] Mafra D, Guebre-Egziabher F, Cleaud C, Arkouche W, Mialon A, Drai J, Fouque D. Obestatin and ghrelin interplay in hemodialysis patients. Nutrition. 2010 Nov-Dec;26(11-12):1100-4. doi: 10.1016/j.nut.2009.09.003. Epub 2009 Dec 16. PMID 20018486
- [Background] Buscher AK, Buscher R, Hauffa BP, Hoyer PF. Alterations in appetite-regulating hormones influence protein-energy wasting in pediatric patients with chronic kidney disease. Pediatr Nephrol. 2010 Nov;25(11):2295-301. doi: 10.1007/s00467-010-1588-9. Epub 2010 Jul 6. PMID 20607302
- [Background] Nusken KD, Groschl M, Rauh M, Stohr W, Rascher W, Dotsch J. Effect of renal failure and dialysis on circulating ghrelin concentration in children. Nephrol Dial Transplant. 2004 Aug;19(8):2156-7. doi: 10.1093/ndt/gfh310. No abstract available. PMID 15252183
- [Background] Arbeiter AK, Buscher R, Petersenn S, Hauffa BP, Mann K, Hoyer PF. Ghrelin and other appetite-regulating hormones in paediatric patients with chronic renal failure during dialysis and following kidney transplantation. Nephrol Dial Transplant. 2009 Feb;24(2):643-6. doi: 10.1093/ndt/gfn529. Epub 2008 Sep 22. PMID 18809976
- [Derived] Monzani A, Perrone M, Prodam F, Moia S, Genoni G, Testa S, Paglialonga F, Rapa A, Bona G, Montini G, Edefonti A. Unacylated ghrelin and obestatin: promising biomarkers of protein energy wasting in children with chronic kidney disease. Pediatr Nephrol. 2018 Apr;33(4):661-672. doi: 10.1007/s00467-017-3840-z. Epub 2017 Nov 18. PMID 29150712